CLINICAL TRIAL: NCT01928147
Title: A Phase Ia and Ib Dose-Ranging Study to Assess the Safety, Pharmacokinetics, and Antiviral Efficacy of PPI-383 in Healthy Adults and Hepatitis C Patients
Brief Title: A Phase 1a/1b Study of PPI-383 in Healthy Adults and Hepatitis C Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Presidio Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPI-383-101
Record Dates: First submitted 2013-08-19; First posted 2013-08-23 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C, Chronic
Keywords: NS5B polymerase inhibitor; Phase 1; Genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PPI-383 single dose escalation in healthy volunteers (Experimental): There will be up to 10 sequential single dose cohorts to assess the bioavailability of different doses and formulations; a food effect cohort will be included.
  Interventions: Drug: PPI-383; Drug: Placebo
- PPI-383 multiple doses in healthy volunteers (Experimental): Upon completion of the single dose cohorts, an additional cohort will receive the highest well-tolerated dose from the single dose cohorts or placebo once daily for five days; up to additional cohorts may receive multiple doses of different formulations or different regimens
  Interventions: Drug: PPI-383; Drug: Placebo
- PPI-383 multiple dose escalation in HCV Subjects (Experimental): Upon completion of the single and multiple dose healthy volunteer cohorts, there will be 3, and potentially 4, sequential cohorts of HCV patients
  Interventions: Drug: PPI-383; Drug: Placebo

INTERVENTIONS:
Drug: PPI-383
Drug: Placebo

SUMMARY:
PPI-383 is an antiviral agent (an inhibitor of the hepatitis C virus NS5B polymerase) that is being developed as a potential treatment for hepatitis C virus infection. This study is being done to assess the dose-related safety and tolerance of PPI-383 when given to healthy volunteers for up to 5 days (Part I of the study) and to hepatitis C patients for up to 3 days (Part II). In addition, the study will assess how much PPI-383 is absorbed into the bloodstream. In Part II, the dose-related effect of PPI-383 on the amount of hepatitis C virus in patients' bloodstream (serum HCV RNA levels) also will be assessed.

ELIGIBILITY:
Part I volunteers (single and multiple dose) - key inclusion criteria

* Healthy males
* Age 18 to 55 years
* Body mass index (BMI)18 to 32 kg/m2

Part II patients- key inclusion criteria

* Males, or females of non-childbearing potential
* Age 18 to 65 years
* Chronic hepatitis C, and absence of other known liver disease
* Seropositive for HCV antibody (HCV Ab) or HCV RNA at least once previously
* Seropositive for HCV Ab at screening
* Serum HCV RNA > 5 log10 IU/mL at screening
* HCV gt-1
* Treatment-naïve for hepatitis C:
* BMI 18 to 35 kg/m2
* Otherwise in good health, without severe or clinically significant chronic or recurrent conditions requiring frequent medical intervention or continual pharmacologic management, except for anti-hypertensive use
* No medical or psychosocial conditions that would potentially interfere with the subject's ability to comply with the study assessments or visit schedule.

Part II patients - key exclusion criteria

* Seropositive for human immunodeficiency virus (HIV) antibody or hepatitis B virus (HBV) surface antigen (HBsAg)
* Signs or symptoms of decompensated liver disease
* Evidence of cirrhosis or hepatocellular carcinoma
* Diabetes Mellitus treated with insulin or hypoglycemic agents
* Asthma requiring hospital admission within the preceding 12 months
* History of alcohol abuse or illicit drug use which could interfere with a patient's compliance with the protocol requirements
* Any of the following laboratory values at screening

  * Haemoglobin (Hgb) <11 g/dL in women or 12 g/dL in men
  * White blood cell count <4,000/mm3
  * Absolute neutrophil count (ANC) < 1800 per mm3
  * Platelet count <100,000 per mm3
  * Serum creatinine > upper limit of normal (ULN) at the central study laboratory
  * Serum albumin <3.4 g/dL
  * Total bilirubin >2.0 mg/dL
* Clinically significant abnormality in the electrocardiograms (ECGs) at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as measured by clinical adverse events and laboratory assessments | Part I, up to day 12; and Part II, up to day 17

SECONDARY OUTCOMES:
PPI-383 plasma levels | Part I, up to day 12; and Part II, up to day 17
serum HCV RNA levels | Part II, up to day 17

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Brown, M.D., Study Director — Presidio Pharmaceuticals
Locations (3):
- Investigational site, Phoenix, Mauritius
- United Kingdom (2):
  - Investigational site, London
  - Investigational site, Nottingham